CLINICAL TRIAL: NCT01980095
Title: A Randomized Placebo-Controlled Phase 3 Study to Assess the Safety and Efficacy of RHB-105 in the Treatment of Confirmed Helicobacter Pylori (H. Pylori) Infection in Non-investigated Dyspepsia Patients
Brief Title: ERADICATE Hp - Treating Helicobacter Pylori With RHB-105
Acronym: ERADICATE Hp
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RHB-105-01
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Dyspepsia; Helicobacter Pylori Infection
Keywords: Helicobacter pylori; H. pylori; Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RHB-105 (Experimental): RHB-105 is an 'all-in-one' combination oral capsule consisting of 2 different antibiotics and a proton pump inhibitor combined in a single capsule.
  Interventions: Drug: RHB-105
- Placebo (Placebo Comparator): Capsules that look like the RHB-105 product but contain no active ingredient.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RHB-105 — The intended dose is RHB-105 (12.5 mg rifabutin, 250 mg amoxicillin, and 10 mg omeprazole capsules) 4 capsules every eight hours, equivalent to a total daily dose of:
  * Rifabutin 150 mg
  * Amoxicillin 3000 mg
  * Omeprazole 120 mg
  Subjects will take study drug every 8 hours with food for 14 consecutive days.
  Arms: RHB-105
Drug: Placebo — Subjects will take 4 placebo capsules every 8 hours with food for 14 days.
  Arms: Placebo

SUMMARY:
The "test and treat" strategy for treating dyspeptic patients who are H. pylori positive is rapidly becoming the standard of care. This study will test the effectiveness of RHB-105, a new triple therapy to treat H. pylori infection in dyspeptic patients.

DETAILED DESCRIPTION:
This is a, randomized, double-blind, placebo-controlled study of RHB-105 in adult subjects complaining of epigastric discomfort that have been screened and found to be positive for H. pylori infection via 13C Urea Breath Test (UBT) and either fecal antigen test or CLO test.

Eligible subjects will be randomized in a ratio of 1:2 between placebo arm (n=30) and the active arm (RHB-105) (n=60). Subjects will receive study drug for 14 consecutive days. Eradication of H. pylori infection will be determined based on 13C UBT conducted between 28 to 56 days after completion of study drug therapy.

Subjects will be unblinded upon 13C UBT analysis. This will provide timely active therapy to all subjects enrolled in this study. Subjects in the placebo arm will be entitled to receive standard-of-care as prescribed by the treating physician following un-blinding.

Eradication failures (13C UBT-positive) in the active study drug arm will undergo upper endoscopy with sampling for culture and sensitivity testing (to rifabutin, amoxicillin, clarithromycin, and metronidazole). Culture and sensitivity directed therapy as prescribed by the treating physician will be offered to these subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age and ≤ 65 years
2. Have symptoms consistent with dyspepsia of at least two weeks duration (defined as recurrent pain or discomfort centered in the upper abdomen, often with a relation to meals)
3. Be positive for H. pylori by 13C Urea Breath Test (UBT) and also by fecal antigen test
4. Be informed of the nature of the study and provide written informed consent before any study specific procedures are performed (or have a legally authorized representative sign consent)

Exclusion Criteria:

1. Have alarm symptoms/signs (including unexplained anemia [iron deficiency), melena / hematemesis, anorexia, dysphagia, jaundice, weight loss)
2. Have taken antibiotics in the 4 weeks prior to screening
3. Have taken bismuth containing medications such as peptobismol in the 4 weeks prior to screening
4. Have a history of any previous esophageal or gastric surgery, except for simple closure of perforated ulcer
5. Have a history of gastric outlet obstruction
6. Have a history of hypersecretory state such as Zollinger-Ellison Syndrome
7. Have a history of gastric cancer
8. Have the presence of active gastric and duodenal ulcers or presence of 3 or more active ulcers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Y Graham, MD, Principal Investigator — Baylor College of Medicine
Locations (12):
- United States (12):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Anaheim Clinical Trials, Anaheim, California
  - Catalina Research Institute, Chino, California
  - Jupiter Research, Inc., Jupiter, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - MedPharmics, Metairie, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - MGG Group Co. Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Office of Dr. Stephen Miller, MD, Las Vegas, Nevada
  - Peters Medical Research, High Point, North Carolina
  - Wake Research Associates, Raleigh, North Carolina

REFERENCES:
- [Derived] Howden CW, Sheldon KL, Almenoff JS, Chey WD. Pitfalls of Physician-Directed Treatment of Helicobacter pylori: Results from Two Phase 3 Clinical Trials and Real-World Prescribing Data. Dig Dis Sci. 2022 Sep;67(9):4382-4386. doi: 10.1007/s10620-021-07323-5. Epub 2021 Dec 4. PMID 34862940

RESULTS

PARTICIPANT FLOW:
Groups:
- RHB-105: RHB-105 is an 'all-in-one' combination oral capsule consisting of 2 different antibiotics and a proton pump inhibitor combined in a single capsule.
  Total daily dose of: Rifabutin 150 mg, Amoxicillin 3000 mg and Omeprazole 120 mg
Period: Overall Study
Arm/Group | RHB-105 | Placebo
Started | 78 (Protocol planned for 90 patients, protocol amendment increase up to 120 patients.) | 41 (Protocol planned for 90 patients, protocol amendment increase up to 120 patients.)
Treated | 77 (Of 78 patients randomized, 1 patient erroneously randomized and not treated) | 41
Completed | 63 | 30
Not Completed | 15 | 11
Not completed — Lost to Follow-up | 6 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Poor compliance | 5 | 0
Not completed — Safety issue | 0 | 1
Not completed — Study drug discontinued | 1 | 0
Not completed — Randomized by mistake | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RHB-105 | Placebo | Total
Number analyzed (Participants) | 77 | 41 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (10.56) | 45.8 (9.52) | 46 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 16 | 44
  Male | 49 | 25 | 74

OUTCOME MEASURES:

1. Primary Outcome: The Occurrence of H. Pylori Eradication as Confirmed Via 13C UBT Testing
Description: Modified intent-to-treat (mITT) population analyzed included all participants whok received at least 1 dose of study drug and underwent a 13C Urea Breath Test (UBT) at Visit 4. Participants with negative test results were to be considered treatment successes. Patients who tested positive for H. pylori infection, and those with indeterminate, not assessable, or missing results were to be considered treatment failures. The statistical hypothesis that the active treatment is superior to 70% was to be tested against the alternative hypothesis that the active treatment is statistically indistinguishable or less than 70% effective using a one-sample Z-test.
Time Frame: 28-56 days after completion of treatment
Population: The mITT Population included all subjects who received at least 1 dose of randomized study treatment and underwent a 13C UBT test at Visit 4. This population consisted in 66 subjects in the RHB-105 group and 37 subjects in the placebo group.
Measure: Count of Participants; unit: Participants
Groups:
- RHB-105: RHB-105 is an 'all-in-one' combination oral capsule consisting of 2 different antibiotics and a proton pump inhibitor combined in a single capsule.
  Total daily dose of:
  * Rifabutin 150 mg
  * Amoxicillin 3000 mg
  * Omeprazole 120 mg
Arm/Group | RHB-105 | Placebo
Number analyzed (Participants) | 66 | 37
Participants
  H. pylori eradication success | 59 | 1
  H. pylori eradication failure | 7 | 36
Statistical Analysis 1: Comparison: RHB-105; Test type: Superiority or Other; p = 0.001, One-sample Z-test, RHB-105 subjects only

2. Other Pre Specified Outcome: H. Pylori Eradication
Description: The occurrence of H. pylori eradication in Placebo and Active Drug Eradication Failure Patients treated with Standard of Care (SOC) treatment
Time Frame: 28-56 days after completion of SOC treatment
Population: Eradication Failure Subjects at Visit 4 were treated with standard of care therapy by the investigator and performed a 13C Urea Breath Test at Visit 8 to confirm H. pylori eradication. This population included 27 subjects in the placebo group and 4 subjects in the active drug eradication failure subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Subjects: These patients failed h.pylori eradication on study drug (placebo) and were subsequently treated with standard of care therapy as per the investigator
- Active Drug Eradication Failure Subjects: These patients failed h.pylori eradication on study drug (active) and were subsequently treated with standard of care therapy as per the investigator.
Arm/Group | Placebo Subjects | Active Drug Eradication Failure Subjects
Number analyzed (Participants) | 27 | 4
Participants
  H. pylori eradication success | 17 | 2
  H. pylori eradication failure | 10 | 2

ADVERSE EVENTS:
Time Frame: 1 year and 10 months
Groups:
- Placebo: Identical capsules that look like the RHB-105 product but contain no active ingredient.
Arm/Group | RHB-105 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/77 | 1/41
Other Adverse Events (participants affected / at risk) | 38/77 | 17/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHB-105 (N=77) | Placebo (N=41)
Anemia of Grade 3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Perirectal Abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHB-105 (N=77) | Placebo (N=41)
Diarrhoea (Gastrointestinal disorders) | 11 (14) | 4 (4)
Abdominal tenderness (Gastrointestinal disorders) | 5 (5) | 3 (3)
Flatulence (Gastrointestinal disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 10 (13) | 4 (4)
Dizziness (Nervous system disorders) | 3 (4) | 3 (3)
Chromaturia (Renal and urinary disorders) | 10 (10) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agree that the Sponsor shall have the right to the first publication of the results of the Study. Following the first publication, the PI may publish data or results from the Study; subject to Sponsor for review and approval in writing at least sixty (60) days prior to the date of the publication. Sponsor may require changes and may extend the embargo to protect its intellectual property or other proprietary interests and to allow for the taking actions for this purpose.